CLINICAL TRIAL: NCT05811325
Title: Effect of Kinesio Taping With and Without Craniosacral Therapy on Pain, Disability, and Quality of Life in Pregnent Female With Sacroiliac Joint Dysfunction
Brief Title: Kinesio Taping With &Without Craniosacral Therapy in Pregnant Females With SIJ Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0538
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Sacral Disorder
Keywords: Sacro-iliac dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio taping without craniosacral therapy (Experimental): This group received Kinesio taping for improvement in pain,disability and quality of life.
  Interventions: Other: kinesiotaping without craniosacral therapy
- kinesio taping group with craniosacral therapy (Active Comparator): Group received kinesio Taping with craniosacral therapy for improvement in pain,disability and quality of life.
  Interventions: Other: kinesiotaping with craniosacral therapy

INTERVENTIONS:
Other: kinesiotaping without craniosacral therapy — The first treatment group will receive kinesio taping for 6 weeks atleast 4 times per week
  Arms: kinesio taping without craniosacral therapy
Other: kinesiotaping with craniosacral therapy — The second treatment group will receive kinesio taping with craniosacral therapy for 6 weeks atleast 4 times per week with each session lasting for 60 minutes
  Arms: kinesio taping group with craniosacral therapy

SUMMARY:
SIJ dysfunction adversely affects quality of life and causes functional impairment and disability. Although, K taping and craniosacral therapy were previously affective in treating SI joint dysfunction, the combined affects of these intervention have not been compared previously to K taping alone.

DETAILED DESCRIPTION:
This study is a randomized controlled trial and have 30 pregnant women suffering from SIJH dysfunction. There is 2 groups and both have received treatment for 6 weeks. The data on pain is collected through VAS and the data on disability is collected through Oswestry Disability Index, and data on quality of life will be collected using SF-36. Measurements will be taken at the beginning of the study and at the end of the 4th week, at the completion of the study. Data will be analyzed using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-35
* pregnant females in 3rd trimester
* pregnant females with SIJ dysfunction

Exclusion Criteria:

* high risk pregnancy
* pregnant females with hypermobility syndrome
* previous pelvic history

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnent females
Enrollment: 30 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
VISUAL ANALOGUE SCALE | 6 WEEKS
  This scale is used to assess pain.
Oswestry Disability Index | 4 weeks
  it is used to measure disability.

SECONDARY OUTCOMES:
SF-36 | 4 weeks
  Data on quality of life is measured by this scale.

CONTACTS AND LOCATIONS:
Overall Officials: tahreem Masood, Principal Investigator — ripah international university
Locations (1):
- Mayo Hopital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No